CLINICAL TRIAL: NCT00640666
Title: Changes in Cancer-related Cytokines After Participation in a Physical Activity Behavior Change Intervention (CICK Study)
Acronym: CICK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ROG-SIU.003
Record Dates: First submitted 2008-03-13; First posted 2008-03-21 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Exercise; Biomarkers
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity intervention (Experimental): Behavior change intervention
  Interventions: Behavioral: Exercise Behavior Change
- Standard of care with written materials (No Intervention): Written materials

INTERVENTIONS:
Behavioral: Exercise Behavior Change — Multidisciplinary
  Other Names: physical activity; exercise
  Arms: Physical activity intervention

SUMMARY:
It is important to confirm health benefits experienced by breast cancer survivors after participation in a physical activity behavior change intervention. One such potential benefit is a reduction in harmful inflammation that might lead to increased symptoms or cancer risk. Because little is known about how physical activity behavior change interventions influence inflammation in breast cancer survivors, the investigators study will measure inflammation with blood markers known as cytokines among breast cancer survivors before and after a physical activity intervention. Such information has the potential to lead to improved physical functioning, reduction in bothersome symptoms (e.g., fatigue), and reduced cancer risk in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients between the ages of 18 and 70 years of age with a diagnosis of Stage I, II, or IIIA breast cancer who are not currently receiving (and do not plan to receive during the study duration) chemotherapy or radiation therapy. The participant may be taking longer term therapies such as aromatase inhibitors, estrogen receptor modulators, etc.
* If the patient has undergone a surgical procedure, must be at least 8 weeks post-procedure.
* English speaking.
* Medical clearance for participation provided by primary care physician or oncologist.

Exclusion Criteria:

* Diagnosis of dementia or organic brain syndrome.
* Medical, psychological, or social characteristic that would interfere with ability to fully participate in program activities and assessments (e.g., psychosis, schizophrenia, etc.).
* Contraindication to participation in a regular physical activity program.
* Metastatic or recurrent disease
* Inability to ambulate
* Engaged in ≥ 60 minutes of vigorous physical activity or ≥ 150 minutes of moderate plus vigorous activity per week during the past month.
* Anticipates undergoing elective surgery during the duration of the intervention which would interfere with intervention participation (e.g., breast reconstructive surgery).
* Participant does not live or work within 50 miles of the study site.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2013-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in pro-inflammatory and anti-inflammatory cytokines | baseline and 3 months

SECONDARY OUTCOMES:
Change in fatigue, sleep and muscle strength | baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q Rogers, M.D., M.P.H., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Rogers LQ, Markwell SJ, Courneya KS, McAuley E, Verhulst S. Physical activity type and intensity among rural breast cancer survivors: patterns and associations with fatigue and depressive symptoms. J Cancer Surviv. 2011 Mar;5(1):54-61. doi: 10.1007/s11764-010-0160-8. Epub 2010 Nov 26. PMID 21110134
- [Background] Rogers LQ, Vicari S, Courneya KS. Lessons learned in the trenches: facilitating exercise adherence among breast cancer survivors in a group setting. Cancer Nurs. 2010 Nov-Dec;33(6):E10-7. doi: 10.1097/NCC.0b013e3181db699d. PMID 20562618
- [Background] Rogers LQ, Hopkins-Price P, Vicari S, Markwell S, Pamenter R, Courneya KS, Hoelzer K, Naritoku C, Edson B, Jones L, Dunnington G, Verhulst S. Physical activity and health outcomes three months after completing a physical activity behavior change intervention: persistent and delayed effects. Cancer Epidemiol Biomarkers Prev. 2009 May;18(5):1410-8. doi: 10.1158/1055-9965.EPI-08-1045. Epub 2009 Apr 21. PMID 19383889
- [Result] Rogers LQ, Fogleman A, Trammell R, Hopkins-Price P, Vicari S, Rao K, Edson B, Verhulst S, Courneya KS, Hoelzer K. Effects of a physical activity behavior change intervention on inflammation and related health outcomes in breast cancer survivors: pilot randomized trial. Integr Cancer Ther. 2013 Jul;12(4):323-35. doi: 10.1177/1534735412449687. Epub 2012 Jul 24. PMID 22831916
- See also: National Cancer Institute site on Physical Activity and Cancer — http://www.cancer.gov/cancertopics/factsheet/physical-activity-qa